CLINICAL TRIAL: NCT06815497
Title: Phase II Non-Randomized, Unblinded, Single-Center Trial of Telmisartan in Combination With Cytotoxic Regimens in Platinum-Resistant Ovarian Cancer Versus Historical Best Supportive Care
Brief Title: Telmisartan in Combination With Cytotoxic Regimens in Platinum-Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tyler J Curiel (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor-Investigator, Tyler J Curiel, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002599; 24WIL599 (Other: DHMC)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Telmisartan with Standard of Care Treatment (Experimental): oral telmisartan in combination with standard of care chemotherapy. chemotherapy regimen is preferably doxorubicin (preferably liposomal doxorubicin) but paclitaxel, nab-paclitaxel, or docetaxel are allowed per investigator or patient preference
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan — Telmisartan will be introduced as a 40 mg tablet to be taken orally once daily. In participants not experiencing telmisartan dose limiting toxicity, the dose will be escalated to a maximum of 80 mg
  Other Names: Micardis

SUMMARY:
The primary study objective is to assess progression-free survival in patients with ovarian cancer receiving telmisartan plus selected standard of care chemotherapy regimens versus historical controls.

DETAILED DESCRIPTION:
This is an open label, single-arm Phase II trial of telmisartan plus selected standard of care chemotherapy regimens containing an anthracycline or taxane. The primary study objective is to assess progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Able and willing to provide informed consent.
* Histologically proven high-grade serous ovarian carcinomas (HGSOC)
* Platinum-resistant or refractory ovarian cancer (OC) defined as progression of disease on carboplatin or growth of disease as detected on computed tomography (CT) scan within 6 months of last platinum treatment
* To receive the allowable standard of care (SOC) chemotherapy regimens for OC
* Life expectancy ≥2 months
* Adequate organ and bone marrow reserve function as indicated by the following:
* Adequate hematological function, defined as absolute neutrophil count (ANC) ≥1.5 x 10^9/L, platelet count ≥100 x 10^9/L, and hemoglobin ≥8 g/dL without recent transfusion (defined as a transfusion that has occurred within 2 weeks of the hemoglobin measurement)
* Adequate liver function, defined as total bilirubin level ≥1.5 x institutional upper limit of normal (IULN), aspartate aminotransferase (AST) ≤ 2.5 x IULN, and alanine aminotransferase (ALT) ≤ 2.5 x IULN
* Adequate renal function defined as creatinine ≤ 1.5 x IULN or measured or calculated creatinine clearance ≥ 40 mL/min per institutional standard. Assessment methods must be recorded.
* Adequate coagulation, defined as international normalized ratio (INR) or prothrombin time ≤ 1.5 x IULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x IULN (unless patient receiving anticoagulant therapy).
* Female patients of childbearing potential (FCBP) must agree to use highly effective contraceptive method(s) while on this study and for at least 3 months after the last dose of chemotherapy
* FCBP must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Non-childbearing potential is defined as 1 of the following:
* ≥ 45 years of age and has not had menses for >1 year
* Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation
* Status is post-hysterectomy, -oophorectomy, or -tubal ligation
* Genetic defect precluding pregnancy
* No contraindication to telmisartan*, including angiotensin converting enzyme (ACE) inhibitor use in the 6 weeks prior to telmisartan start on trial
* Systolic blood pressure maintained at ≥ 110 mm Hg during study enrollment assessment and throughout the study.

Exclusion Criteria:

Patients who meet any of the criteria below may NOT be eligible to participate in this study:

* Patients who are unable to provide informed consent.
* Patients with known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they must have an undetectable HCV viral load
* Hypertensive urgency or emergency as defined
* Incarcerated or homeless
* Pregnant or lactating.
* Individuals who are not yet adults <18 years of age.
* On lithium therapy in any form
* Received rituximab or amifostine within 30 days prior to first telmisartan dose on this study
* Active, serious infection requiring treatment
* Clinically significant (i.e., active) cardiovascular disease, cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication
* History or current evidence of any condition, therapy, and active infections, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Taking ramapril
* Using bevacizumab as part of their SOC chemotherapy regimen
* If known to be HIV-infected, have undetectable HIV viral load by any accepted standard of care HIV detection method

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 48 months
  Progression free survival is defined as the time between the initiation of telmisartan to progression, as defined by RECIST criteria, on a computed tomography scan.

SECONDARY OUTCOMES:
Treatment tolerability | 24 months
  Treatment tolerability will be quantified as the proportion of patients with a toxicity related to telmisartan and the proportion of patients who stopped telmisartan due to its toxicity
Circulating tumor DNA changes | 24 months
  Peripheral blood will be drawn throughout the study and tested for circulating tumor DNA (ctDNA) damage. The goal is to understand tumor genetic changes in response to adding telmisartan to test if changes predictive of treatment response or failure can be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Wilkinson-Ryan, MD, Principal Investigator — Dartmouth Health
Locations (2):
- United States (2):
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Dartmouth-Hitchcock Manchester, Manchester, New Hampshire

REFERENCES:
- [Background] Richardson DL, Eskander RN, O'Malley DM. Advances in Ovarian Cancer Care and Unmet Treatment Needs for Patients With Platinum Resistance: A Narrative Review. JAMA Oncol. 2023 Jun 1;9(6):851-859. doi: 10.1001/jamaoncol.2023.0197. PMID 37079311
- [Background] Moore KN, Angelergues A, Konecny GE, Garcia Y, Banerjee S, Lorusso D, Lee JY, Moroney JW, Colombo N, Roszak A, Tromp J, Myers T, Lee JW, Beiner M, Cosgrove CM, Cibula D, Martin LP, Sabatier R, Buscema J, Estevez-Garcia P, Coffman L, Nicum S, Duska LR, Pignata S, Galvez F, Wang Y, Method M, Berkenblit A, Bello Roufai D, Van Gorp T; Gynecologic Oncology Group Partners and the European Network of Gynaecological Oncological Trial Groups. Mirvetuximab Soravtansine in FRalpha-Positive, Platinum-Resistant Ovarian Cancer. N Engl J Med. 2023 Dec 7;389(23):2162-2174. doi: 10.1056/NEJMoa2309169. PMID 38055253
- [Background] Mellman I, Chen DS, Powles T, Turley SJ. The cancer-immunity cycle: Indication, genotype, and immunotype. Immunity. 2023 Oct 10;56(10):2188-2205. doi: 10.1016/j.immuni.2023.09.011. PMID 37820582
- [Background] Drerup JM, Liu Y, Padron AS, Murthy K, Hurez V, Zhang B, Curiel TJ. Immunotherapy for ovarian cancer. Curr Treat Options Oncol. 2015 Jan;16(1):317. doi: 10.1007/s11864-014-0317-1. PMID 25648541
- [Background] Palaia I, Tomao F, Sassu CM, Musacchio L, Benedetti Panici P. Immunotherapy For Ovarian Cancer: Recent Advances And Combination Therapeutic Approaches. Onco Targets Ther. 2020 Jun 26;13:6109-6129. doi: 10.2147/OTT.S205950. eCollection 2020. PMID 32617007
- [Background] Muaibati M, Abuduyilimu A, Zhang T, Dai Y, Li R, Huang F, Li K, Tong Q, Huang X, Zhuang L. Efficacy of immune checkpoint inhibitor monotherapy or combined with other small molecule-targeted agents in ovarian cancer. Expert Rev Mol Med. 2023 Jan 24;25:e6. doi: 10.1017/erm.2023.3. PMID 36691778
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Zhang L, Conejo-Garcia JR, Katsaros D, Gimotty PA, Massobrio M, Regnani G, Makrigiannakis A, Gray H, Schlienger K, Liebman MN, Rubin SC, Coukos G. Intratumoral T cells, recurrence, and survival in epithelial ovarian cancer. N Engl J Med. 2003 Jan 16;348(3):203-13. doi: 10.1056/NEJMoa020177. PMID 12529460
- [Background] Curiel TJ, Coukos G, Zou L, Alvarez X, Cheng P, Mottram P, Evdemon-Hogan M, Conejo-Garcia JR, Zhang L, Burow M, Zhu Y, Wei S, Kryczek I, Daniel B, Gordon A, Myers L, Lackner A, Disis ML, Knutson KL, Chen L, Zou W. Specific recruitment of regulatory T cells in ovarian carcinoma fosters immune privilege and predicts reduced survival. Nat Med. 2004 Sep;10(9):942-9. doi: 10.1038/nm1093. Epub 2004 Aug 22. PMID 15322536
- [Background] Mariniello M, Petruzzelli R, Wanderlingh LG, La Montagna R, Carissimo A, Pane F, Amoresano A, Ilyechova EY, Galagudza MM, Catalano F, Crispino R, Puchkova LV, Medina DL, Polishchuk RS. Synthetic Lethality Screening Identifies FDA-Approved Drugs that Overcome ATP7B-Mediated Tolerance of Tumor Cells to Cisplatin. Cancers (Basel). 2020 Mar 6;12(3):608. doi: 10.3390/cancers12030608. PMID 32155756
- [Background] Fujita N, Fujita K, Iwama H, Kobara H, Fujihara S, Chiyo T, Namima D, Yamana H, Kono T, Takuma K, Hirata M, Kobayashi K, Kato K, Kamada H, Morishita A, Tsutsui K, Himoto T, Okano K, Suzuki Y, Masaki T. Antihypertensive drug telmisartan suppresses the proliferation of gastric cancer cells in vitro and in vivo. Oncol Rep. 2020 Jul;44(1):339-348. doi: 10.3892/or.2020.7607. Epub 2020 May 7. PMID 32627043
- [Background] Samukawa E, Fujihara S, Oura K, Iwama H, Yamana Y, Tadokoro T, Chiyo T, Kobayashi K, Morishita A, Nakahara M, Kobara H, Mori H, Okano K, Suzuki Y, Himoto T, Masaki T. Angiotensin receptor blocker telmisartan inhibits cell proliferation and tumor growth of cholangiocarcinoma through cell cycle arrest. Int J Oncol. 2017 Dec;51(6):1674-1684. doi: 10.3892/ijo.2017.4177. Epub 2017 Oct 23. PMID 29075786
- [Background] Oura K, Tadokoro T, Fujihara S, Morishita A, Chiyo T, Samukawa E, Yamana Y, Fujita K, Sakamoto T, Nomura T, Yoneyama H, Kobara H, Mori H, Iwama H, Okano K, Suzuki Y, Masaki T. Telmisartan inhibits hepatocellular carcinoma cell proliferation in vitro by inducing cell cycle arrest. Oncol Rep. 2017 Nov;38(5):2825-2835. doi: 10.3892/or.2017.5977. Epub 2017 Sep 20. PMID 29048654
- [Background] Fujihara S, Morishita A, Ogawa K, Tadokoro T, Chiyo T, Kato K, Kobara H, Mori H, Iwama H, Masaki T. The angiotensin II type 1 receptor antagonist telmisartan inhibits cell proliferation and tumor growth of esophageal adenocarcinoma via the AMPKalpha/mTOR pathway in vitro and in vivo. Oncotarget. 2017 Jan 31;8(5):8536-8549. doi: 10.18632/oncotarget.14345. PMID 28052030
- [Background] Pu Z, Zhu M, Kong F. Telmisartan prevents proliferation and promotes apoptosis of human ovarian cancer cells through upregulating PPARgamma and downregulating MMP-9 expression. Mol Med Rep. 2016 Jan;13(1):555-9. doi: 10.3892/mmr.2015.4512. Epub 2015 Nov 6. PMID 26548340
- [Background] Green R, Howell M, Khalil R, Nair R, Yan J, Foran E, Katiri S, Banerjee J, Singh M, Bharadwaj S, Mohapatra SS, Mohapatra S. Actinomycin D and Telmisartan Combination Targets Lung Cancer Stem Cells Through the Wnt/Beta Catenin Pathway. Sci Rep. 2019 Dec 3;9(1):18177. doi: 10.1038/s41598-019-54266-z. PMID 31796785
- [Background] Rasheduzzaman M, Moon JH, Lee JH, Nazim UM, Park SY. Telmisartan generates ROS-dependent upregulation of death receptor 5 to sensitize TRAIL in lung cancer via inhibition of autophagy flux. Int J Biochem Cell Biol. 2018 Sep;102:20-30. doi: 10.1016/j.biocel.2018.06.006. Epub 2018 Jun 19. PMID 29929000
- [Background] Ozeki K, Tanida S, Morimoto C, Inoue Y, Mizoshita T, Tsukamoto H, Shimura T, Kataoka H, Kamiya T, Nishiwaki E, Ishiguro H, Higashiyama S, Joh T. Telmisartan inhibits cell proliferation by blocking nuclear translocation of ProHB-EGF C-terminal fragment in colon cancer cells. PLoS One. 2013;8(2):e56770. doi: 10.1371/journal.pone.0056770. Epub 2013 Feb 22. PMID 23451083
- [Background] Kobara H, Fujihara S, Iwama H, Matsui T, Fujimori A, Chiyo T, Tingting S, Kobayashi N, Nishiyama N, Yachida T, Tadokoro T, Oura K, Tani J, Fujita K, Nomura T, Yoneyama H, Morishita A, Okano K, Suzuki Y, Mori H, Masaki T. Antihypertensive drug telmisartan inhibits cell proliferation of gastrointestinal stromal tumor cells in vitro. Mol Med Rep. 2020 Aug;22(2):1063-1071. doi: 10.3892/mmr.2020.11144. Epub 2020 May 14. PMID 32626983
- [Background] Uemura H, Ishiguro H, Nakaigawa N, Nagashima Y, Miyoshi Y, Fujinami K, Sakaguchi A, Kubota Y. Angiotensin II receptor blocker shows antiproliferative activity in prostate cancer cells: a possibility of tyrosine kinase inhibitor of growth factor. Mol Cancer Ther. 2003 Nov;2(11):1139-47. PMID 14617787
- [Background] Wu TT, Niu HS, Chen LJ, Cheng JT, Tong YC. Increase of human prostate cancer cell (DU145) apoptosis by telmisartan through PPAR-delta pathway. Eur J Pharmacol. 2016 Mar 15;775:35-42. doi: 10.1016/j.ejphar.2016.02.017. Epub 2016 Feb 4. PMID 26852954
- [Background] Takahashi S, Uemura H, Seeni A, Tang M, Komiya M, Long N, Ishiguro H, Kubota Y, Shirai T. Therapeutic targeting of angiotensin II receptor type 1 to regulate androgen receptor in prostate cancer. Prostate. 2012 Oct 1;72(14):1559-72. doi: 10.1002/pros.22505. Epub 2012 Mar 16. PMID 22430461
- [Background] Koyama N, Nishida Y, Ishii T, Yoshida T, Furukawa Y, Narahara H. Telmisartan induces growth inhibition, DNA double-strand breaks and apoptosis in human endometrial cancer cells. PLoS One. 2014 Mar 25;9(3):e93050. doi: 10.1371/journal.pone.0093050. eCollection 2014. PMID 24667764
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123
- [Background] Waight JD, Chand D, Dietrich S, Gombos R, Horn T, Gonzalez AM, Manrique M, Swiech L, Morin B, Brittsan C, Tanne A, Akpeng B, Croker BA, Buell JS, Stein R, Savitsky DA, Wilson NS. Selective FcgammaR Co-engagement on APCs Modulates the Activity of Therapeutic Antibodies Targeting T Cell Antigens. Cancer Cell. 2018 Jun 11;33(6):1033-1047.e5. doi: 10.1016/j.ccell.2018.05.005. PMID 29894690
- [Background] Jensterle M, Janez A, Vrtovec B, Meden-Vrtovec H, Pfeifer M, Prezelj J, Kocjan T. Decreased androgen levels and improved menstrual pattern after angiotensin II receptor antagonist telmisartan treatment in four hypertensive patients with polycystic ovary syndrome: case series. Croat Med J. 2007 Dec;48(6):864-70. doi: 10.3325/cmj.2007.6.864. PMID 18074422
- [Background] Cernes R, Mashavi M, Zimlichman R. Differential clinical profile of candesartan compared to other angiotensin receptor blockers. Vasc Health Risk Manag. 2011;7:749-59. doi: 10.2147/VHRM.S22591. Epub 2011 Dec 12. PMID 22241949
- [Background] Tascilar K, Azoulay L, Dell'Aniello S, Bartels DB, Suissa S. The Use of Telmisartan and the Incidence of Cancer. Am J Hypertens. 2016 Dec 1;29(12):1358-1365. doi: 10.1093/ajh/hpw095. PMID 27557862
- [Background] McAlister FA; Renin Angiotension System Modulator Meta-Analysis Investigators. Angiotensin-converting enzyme inhibitors or angiotensin receptor blockers are beneficial in normotensive atherosclerotic patients: a collaborative meta-analysis of randomized trials. Eur Heart J. 2012 Feb;33(4):505-14. doi: 10.1093/eurheartj/ehr400. Epub 2011 Oct 31. PMID 22041554
- [Background] Galle J. Reduction of proteinuria with angiotensin receptor blockers. Nat Clin Pract Cardiovasc Med. 2008 Jul;5 Suppl 1:S36-43. doi: 10.1038/ncpcardio0806. PMID 18580865
- [Background] Uemura H, Hasumi H, Kawahara T, Sugiura S, Miyoshi Y, Nakaigawa N, Teranishi J, Noguchi K, Ishiguro H, Kubota Y. Pilot study of angiotensin II receptor blocker in advanced hormone-refractory prostate cancer. Int J Clin Oncol. 2005 Dec;10(6):405-10. doi: 10.1007/s10147-005-0520-y. PMID 16369744
- [Background] Colombo N, Van Gorp T, Matulonis UA, Oaknin A, Grisham RN, Fleming GF, Olawaiye AB, Nguyen DD, Greenstein AE, Custodio JM, Pashova HI, Tudor IC, Lorusso D. Relacorilant + Nab-Paclitaxel in Patients With Recurrent, Platinum-Resistant Ovarian Cancer: A Three-Arm, Randomized, Controlled, Open-Label Phase II Study. J Clin Oncol. 2023 Oct 20;41(30):4779-4789. doi: 10.1200/JCO.22.02624. Epub 2023 Jun 26. PMID 37364223
- [Background] Funao K, Matsuyama M, Kawahito Y, Sano H, Chargui J, Touraine JL, Nakatani T, Yoshimura R. Telmisartan is a potent target for prevention and treatment in human prostate cancer. Oncol Rep. 2008 Aug;20(2):295-300. PMID 18636189
- [Background] Daniel B, Nagy G, Czimmerer Z, Horvath A, Hammers DW, Cuaranta-Monroy I, Poliska S, Tzerpos P, Kolostyak Z, Hays TT, Patsalos A, Houtman R, Sauer S, Francois-Deleuze J, Rastinejad F, Balint BL, Sweeney HL, Nagy L. The Nuclear Receptor PPARgamma Controls Progressive Macrophage Polarization as a Ligand-Insensitive Epigenomic Ratchet of Transcriptional Memory. Immunity. 2018 Oct 16;49(4):615-626.e6. doi: 10.1016/j.immuni.2018.09.005. PMID 30332629
- [Background] Kornepati AVR, Rogers CM, Sung P, Curiel TJ. The complementarity of DDR, nucleic acids and anti-tumour immunity. Nature. 2023 Jul;619(7970):475-486. doi: 10.1038/s41586-023-06069-6. Epub 2023 Jul 19. PMID 37468584
- [Background] Washida K, Ihara M, Nishio K, Fujita Y, Maki T, Yamada M, Takahashi J, Wu X, Kihara T, Ito H, Tomimoto H, Takahashi R. Nonhypotensive dose of telmisartan attenuates cognitive impairment partially due to peroxisome proliferator-activated receptor-gamma activation in mice with chronic cerebral hypoperfusion. Stroke. 2010 Aug;41(8):1798-806. doi: 10.1161/STROKEAHA.110.583948. Epub 2010 Jul 1. PMID 20595663
- [Background] Torika N, Asraf K, Danon A, Apte RN, Fleisher-Berkovich S. Telmisartan Modulates Glial Activation: In Vitro and In Vivo Studies. PLoS One. 2016 May 17;11(5):e0155823. doi: 10.1371/journal.pone.0155823. eCollection 2016. PMID 27187688
- [Background] Wilk M, Wasko-Grabowska A, Skoneczna I, Szmit S. Angiotensin System Inhibitors May Improve Outcomes of Patients With Castration-Resistant Prostate Cancer During Abiraterone Acetate Treatment-A Cardio-Oncology Study. Front Oncol. 2021 Apr 1;11:664741. doi: 10.3389/fonc.2021.664741. eCollection 2021. PMID 33869068
- [Background] Peixoto AJ. Acute Severe Hypertension. N Engl J Med. 2019 Nov 7;381(19):1843-1852. doi: 10.1056/NEJMcp1901117. No abstract available. PMID 31693807
- [Background] Sharma P, Nagarajan V. Q: Can an ARB be given to patients who have had angioedema on an ACE inhibitor? Cleve Clin J Med. 2013 Dec;80(12):755-7. doi: 10.3949/ccjm.80a.13041. No abstract available. PMID 24307158